CLINICAL TRIAL: NCT03676660
Title: The Evaluation of Care Demand and Intervention Models for Individuals With ASD in Taiwan
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201707041RINA
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of autism in Taiwan has been significantly increasing over this decade. Though early intervention program and special and resource education have been applied in helping individuals with autism in Taiwan, studies regarding autism in this country so far focus mostly on the prevalence and demographics in restricted populations, diagnostic category, single case observation, and clinical research. Although the data of needs of care and intervention models in autism emerges in Western countries, there is a lack of such data in Taiwan. Due to the high prevalence, long-term impairing and lack of effective prevention, detection, and treatment for autism, tremendous of the resource is needed to be given to individuals with autism. However, the investigators do not know the gap between the need and provided care in currently. This study aims to understand the current state of needs of care and intervention in autism from different stakeholders to inform and improve the health care policies for autism and to establish a holistic care/intervention model for autism in Taiwan.

DETAILED DESCRIPTION:
This study will enroll individuals with autism and their family members from autism-related medical, nongovernmental organizations, and general educational settings, where from elementary schools to colleges, in Taiwan. For patients and their family, the investigators will enroll total 2000 adult individuals with autism and their family members for the questionnaire survey. The needs of assessment and care, and intervention models in autism will be examined using the Chinese version of Camberwell Assessment of Need, autistic traits assessment, emotional difficulty questionnaire, quality of life and Self-administered questionnaire with different versions for stakeholders. The guides for parents and clinicians on autism will be discussed with the patient and family representatives and developed by different autism stakeholders, experts, and scholars based on regular research meetings. Quantitative analyses will be conducted to understand the need and difficulty of care and interventions in autism across different developmental stage.

The investigators anticipate to find differences in care needs by personal characteristics. The survey of the care needs of autism will provide family members, medical and nursing personnel, and related caregivers more information about understanding their care requirements. These results will help the government for the formulation of policies related to early treatment and long-term care. Finally, the guides for parents and clinician on autism would be suggested references.

ELIGIBILITY:
Inclusion Criteria:

* individuals with autism from autism-related medical, nongovernmental organizations, and general educational settings, where from elementary schools to colleges, in Taiwan.

Exclusion Criteria:

* family members of autism cannot complete questionnaire survey will be excluded from the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: For patients and their family, we will enroll total 2000 adult individuals with autism and their family members for the questionnaire survey. The needs of assessment and care, and intervention models in autism will be examined using the Chinese version of Camberwell Assessment of Need, autistic traits assessment, emotional difficulty questionnaire, quality of life and Self-administered questionnaire with different versions for stakeholders.
Sampling Method: Non-Probability Sample
Enrollment: 1948 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Camberwell Assessment of Need (CAN) | 1 day
  The health and social needs of adults across 22 domains of life, such as accommodation, food, self-care, daytime activities, psychotic symptoms, childcare, money, psychological distress, physical health and relationshipsusing the Chinese version of Camberwell Assessment of Need

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan